CLINICAL TRIAL: NCT05738408
Title: Remote Smoking Cessation in Hospitalized Cardiac Patients: Bridging the Post-discharge
Brief Title: Remote Smoking Cessation in Hospitalized Cardiac Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Sherrie Khadanga, PI, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002035
Record Dates: First submitted 2022-06-06; First posted 2023-02-22 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; secondary prevention
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Usual Care (No Intervention): will receive standard treatment which entails referral to Vermont Quit Network. This network offers a wide range of free cessation services, including NRT and web-based modules on preparing to quit and developing a plan
- Intervention: Financial incentives and nicotine replacement therapy intervention (Experimental): an intervention where patients are assigned to financial incentives and NRT of their choice; use of CO monitor to assess abstinence
  Interventions: Behavioral: Financial Incentives (FI) and Nicotine Replacement Therapy (NRT)

INTERVENTIONS:
Behavioral: Financial Incentives (FI) and Nicotine Replacement Therapy (NRT) — : In the intervention condition, patients will receive both NRT plus a 12-week program of monetary incentives for verified smoking abstinence that will be implemented by our clinic staff
  Arms: Intervention: Financial incentives and nicotine replacement therapy intervention

SUMMARY:
The investigators are proposing to examine new strategies for helping patients hospitalized for an acute coronary event adhere to recommendations to quit smoking. The investigators are interested to see whether offering financial incentives for smoking cessation, combined with medications to ameliorate withdrawal, can significantly reduce smoking in a population for which continued smoking has disproportionately negative health effects. The proposed trial can provide significant knowledge for promoting adherence to smoking cessation guidelines in patients with cardiac disease

DETAILED DESCRIPTION:
Cigarette smoking is the leading cause of preventable death in the U.S. The effect of smoking in those with coronary artery disease (CAD) is particularly powerful given that at hospital admission, 27-36% of these patients are active smokers which is much higher than in the general population (<18%).1-3While smoking rates have declined in the U.S., this has not been observed in cardiac populations. Continued smoking after hospitalization also predicts additional negative outcomes such as lack of engagement in comprehensive secondary prevention for example cardiac rehabilitation (CR).4 Smoking may also directly impede improvements in fitness which is a critical predictor of recovery in this population and thus crucial to examine.5-7 Surprisingly, having a serious cardiac event, such as a myocardial infarction (MI) may not be enough to promote sustained cessation.8 Thus, promoting adherence to smoking cessation guidelines in this population is of utmost importance.9

Acute cardiac hospitalization does provide an ideal opportunity to intervene on smoking.10 Patients are required to abstain from smoking while hospitalized and are often motivated to quit. Unfortunately, less than a quarter of patients receive Nicotine Replacement Therapy (NRT) in-hospital and even fewer receive support after discharge. 11,12 For most patients, follow-up care may not occur for 4-6 weeks and most patients relapse to smoking within the first few weeks.11,13 Ideally, intensive intervention would be started in-hospital and continue after discharge, bridging this post-hospital gap in care.

Financial incentives (FI) for objectively verified smoking abstinence is highly effective in promoting smoking cessation in medically vulnerable populations, but, to the Investigators knowledge, has not been tested in patients with CVD.14.15 NRT is safe in cardiac patients, but is rarely prescribed or offered in a manner that maximizes efficacy (i.e., combination short and long-acting NRT).16 Building on our strong published and preliminary data, the investigators hypothesize that a combined behavioral and pharmacologic smoking cessation intervention started in hospital and continued remotely can bridge the post-hospital care gap and support patients through a critical period in cardiac recovery where risk of smoking relapse is high.

ELIGIBILITY:
Inclusion Criteria:

Patients will be recruited if they:

1. Hospitalization for an acute coronary event which includes myocardial infarction or coronary revascularization (percutaneous intervention or coronary artery bypass)
2. live within 30 miles of UVMMC and are >18 years of age
3. Current cigarette smoker (defined as reporting any use of cigarettes in the week before admission and >5 cigarette/day on average over the past 3 months)

Exclusion Criteria:

Patients will be excluded if they have:

1. severe dementia/Alzheimer's disease
2. an active malignancy, excluding non-melanoma skin cancer or low-grade prostate cancer under active surveillance
3. exercise limiting vascular or neuromuscular disease
4. Non-English Speaking
5. No reliable smart-phone
6. Current, regular use of smokeless tobacco or other form of non-combusted tobacco

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical verification of smoking status | 3 months
  Assess the efficacy of combined FI+NRT vs. UC on biochemically verified smoking abstinence

SECONDARY OUTCOMES:
Cardiovascular Fitness | 3 months
  Determine the effect of smoking status on changes in cardiovascular fitness (VO2peak).

OTHER OUTCOMES:
Smoking Characteristics | 3 months
  Cigarettes per day (CPD) using timeline follow back methods
Smoking Characteristics | 3 months
  Fagerstrom Test for Nicotine Dependence [FTND]
Smoking Characteristics | 3 months
  Heaviness of Smoking Index (HSI)
Smoking Characteristics | 3 months
  and the Minnesota Nicotine Withdrawal Scale
Smoking Status | 3 months
  CO monitoring
Physical Function assessed by MOS SF-36 | 3 months
  The General Health Status MOS SF-36 questionnaire will be administered with special attention to the physical function component score.
Quality of Life assessed by EuroQol questionnaire | 3 months
  EuroQol
Quality of Life assessed by MacNew Cardiac Health questionnaire | 3 months
  disease specific MacNew Cardiac Health Status Questionnaire will be administered
Depression assessed by PHQ-9 questionnaire | 3 months
  mood will be measured using the Patient Health Questionnaire (PHQ-9)
Anxiety assessed by GAD-7 Questionnaire | 3 months
  the General Anxiety Disorder questionnaire (GAD-7)Questionnaire will be administered to assess anxiety
Risk Aversion Assessment | 3 months
Health Care Contacts | 12 months
  Combined measure of number of Emergency Department visits and overnight hospitalizations

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided